CLINICAL TRIAL: NCT04899050
Title: Safety and Efficacy of CBD (Epidiolex) in Idiopathic Generalized Epilepsy With Typical Absence Seizures
Brief Title: Epidiolex in Typical Absence Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Selim Benbadis, Professor of Neurology, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY001072
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Study the Efficacy of Epidiolex for Typical Absence Seizures
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Absence Seizures Treated with Epidiolex (Experimental): This is a pilot, open-label study consisting of a screening period of up to 28 Days, a 4-week dose-titration treatment period to dose of up to 20 mg/kg/day BID of CBD (EPIDIOLEX ), and a 30-day safety follow-up period following the last dose of study medication.
  Interventions: Drug: Cannabidiol (Epidiolex)

INTERVENTIONS:
Drug: Cannabidiol (Epidiolex) — Use of Epidiolex to control absence seizures.

SUMMARY:
This is a Pilot study, open-label study consisting of a screening period of up to 4 weeks, a 4-week dose-titration treatment period to dose of up to 20 mg/kg/day BID of CBD (Epidiolex), and a 30 day safety follow-up period following the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant is willing to sign the informed consent form (ICF) indicating that the subject has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
2. Participant is male or female 6 years of age and older, with diagnosis of uncontrolled Genetic (Idiopathic) Generalized Epilepsy with Typical Absence Seizures.
3. Clinical diagnosis of GGE (including, but not limited to, CAE, JAE, juvenile myoclonic epilepsy, or Jeavons syndrome) with absence seizures consistent with the International League against Epilepsy Revised Classification of Seizures (2017).
4. Absence seizures, by history on average once per hour, persisting despite standard of care (SOC) treatment, defined as treatment with at least 2 AEDs appropriate for the patient's epilepsy syndrome. SOC failure, per investigator discretion, will be defined as insufficient clinical response or intolerable side effects, which precludes use of the appropriate AED.
5. Observation of at least 3 instances of generalized discharges of approximately 2.5 - 4 Hz lasting >2 seconds via 24-hr ambulatory EEG.
6. On stable doses of one or more antiepileptic medication(s) for at least 30 days. If a subject is not on medication, adequate documentation justifying lack of therapy may be acceptable for the subject after Greenwich Biosciences review. Ketogenic, modified Atkins diet (MAD), or low glycemic diet with stable carbohydrate ratio for at least 30 days before screening is an acceptable antiepileptic therapy. Vagal nerve stimulation at stable settings (for at least 30 days before screening), without use of the magnet, is also acceptable.
7. Subjects with reproductive capability, including all males and WOCBP, must agree to practice continuous abstinence or adequate contraception methods (appropriate double barrier method or oral, patch, implant, or injectable contraception) from as soon as feasible during screening period until at least 30 days after the last dose (i.e., intermittent abstinence based on "rhythm," temperature monitoring, or other means of timing is not acceptable). WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy) or is not postmenopausal. Postmenopausal is defined as amenorrhea for ≥12 consecutive months without another cause, and a documented serum follicle stimulating hormone (FSH) level ≥35 mIU/mL.
8. Participants who are able and willing to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Participants will be excluded from the study if any of the following conditions apply:

1. Participant who has history of surgical intervention for treatment of epilepsy.
2. Additional seizure (clinical and electrographic) types, including, but not limited to, epileptic spasms, generalized tonic seizures, atonic seizures, or focal seizures. Subjects with GTCS or myoclonic seizures are eligible for the study.
3. Participants with inadequately treated psychotic or mood disorder (e.g., schizophrenia, major depression, bipolar disorder).
4. Presence of severe intellectual disability, severe autism spectrum disorder, or severe developmental disorder such that the subject cannot sign the ICF or cannot cooperate with the study procedures.
5. Presence of positive urine drug screen for drugs of abuse, except if this is explained by use of an allowed prescription medicine.
6. Significant hepatic (AST/ALT or bilirubin ≥2 × ULN) or renal disease (creatinine clearance ≤39 mL/min).
7. A current C-SSRS score of 4 or 5 at screening or history of suicide attempt within the past year.
8. Participant has any medical condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study.
9. Treatment with an investigational agent within 30 days prior to the first dose of EPIDIOLEX or planning to receive an investigational agent during the study.
10. Concurrent legal use of CBD obtained from a state dispensary.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Amount of epileptiform activity. | From baseline EEG to the EEG after 90 days of treatment.
  The EEG epileptiform activity will be measured in seconds per 24 hours period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No